CLINICAL TRIAL: NCT03962985
Title: Effects of Montreal Museum of Fine Arts Visits and Older Community Dwellers With a Precarious State: An Experimental Study
Brief Title: Effects of Montreal Museum of Fine Arts Visits and Older Community Dwellers With a Precarious State
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Jewish General Hospital (Other)
Responsible Party: Principal Investigator, Olivier Beauchet, MD, Professor of Geriatrics, Jewish General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 2020-1789
Record Dates: First submitted 2019-05-23; First posted 2019-05-24 (Actual); Last update posted 2024-07-23 (Actual); Status verified 2024-07

CONDITIONS: Well Aging; Health Impairment; Social Isolation; Old Age
MeSH Terms: conditions — Social Isolation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Intervention (Other): The 41 participants will attend the guided tours at the Montreal Museum of Fine Arts.
  Interventions: Other: Guided tour at the Montreal Museum of Fine Arts

INTERVENTIONS:
Other: Guided tour at the Montreal Museum of Fine Arts — * The duration of the participation -3 months
  * The duration of the guided tour-45 minutes, each week
  * All participants will be asked to fill out some specific online questionnaires during their participations in the study

SUMMARY:
This study evaluates the effects of MMFA visits on psychological, health, social conditions and personal interactions in older community dwellers with a precarious state and to determine whether these effects may change precarity.

DETAILED DESCRIPTION:
Precarity is a vulnerable state exposing individuals to adverse health, psychological social events. Older adults are exposed to precarity, especially those who were the old generation of immigrants in Canada. Art-based activities have also been proposed to community dwellers and have shown positive effects on health outcomes and are determinants for well-being with aging. The effects of participatory art-based activities on precarity in older adults have never been examined. Recently, the Montreal Museum of Fine Arts (MMFA) developed a new participatory art-based activity which is a 3 month-period of weekly museum visits for precarious populations.

ELIGIBILITY:
Inclusion Criteria:

* Being 65 years and over;
* Precarious condition defined with a score ≥30 (/100)
* Having an Internet access with an electronic device (i.e.; laptop, computer, smartphone, tablet) as the repetitive assessments for this study will be performed on the web platform of the Centre of Excellence on Longevity of McGill University;
* Understanding and writing the different languages of the recruitment centre (i.e., French, English, Chinese.);
* Severe frail condition determined with the Centre of Excellence self-administered questionnaire (CESAM)
* Living in Montreal

Exclusion Criteria:

* A concomitant participation to another clinical trial;
* Participation in another art-based activity;
* Palliative care;
* Living in residence;
* Having a moderate to severe mobility impairment (i.e. using a walker, a wheelchair or being unable to walk alone 10m).

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 41 (Actual)
Dates: Start 2019-07-23 (Actual); Primary Completion 2022-06-01 (Actual); Study Completion 2024-07-01 (Actual)

PRIMARY OUTCOMES:
Precarious social conditions | 3 months
  It will be used a questionnaire called: Evaluation of Health Precariousness and Inequalities in Health Examination Centers(EPICE). This questionnaire has 11 questions that summarize 90% a precarious state. The answer to each question is assigned a coefficient, the sum of the 11 answers gives the EPICES score. The score is continuous and ranges from 0 (no precarious social conditions) to 100 (maximum level of precarious conditions).The threshold of 30 defined a precarious state.

SECONDARY OUTCOMES:
Well-being | 3 months
  It will be used a questionnaire called: Warwick-Edinburgh Mental Well-being Scale questionnaire (WEMWBS).The Warwick-Edinburgh Mental Well-being Scale questionnaire is a validated questionnaire composed by 14 positively worded item scale with five response categories. It covers most aspects of positive mental health (positive thoughts and feelings).

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Beauchet, MD, Principal Investigator — Jewish General Hospital
Locations (1):
- Jewish General Hospital, Montreal, Quebec, Canada